CLINICAL TRIAL: NCT02229994
Title: Development of a New Tool for Dyspnea Measurement (DYSLIM for Dyspnea Limitation) in Chronic Respiratory Diseases
Brief Title: Development of a New Tool for Dyspnea Measurement in Chronic Respiratory Diseases
Acronym: DYSLIM
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Pr Joel COSTE, Hôpital Hôtel Dieu - Unité de Bio Statistiques et Epidémiologiques, Paris (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: 2009-A00181-56
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: COPD (With - Without Rehabilitation); Diffuse Interstitial Lung Diseases; Pulmonary Arterial Hypertension Primary or Secondary (Post Embolic .....); Cystic Fibrosis of the Adult
Keywords: Dyspnea; Self-administered questionnaire; Chronic respiratory disease; COPD; Diffuse interstitial lung diseases; Pulmonary arterial hypertension; Cystic fibrosis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Neoplasm Metastasis; Dyspnea; Pulmonary Arterial Hypertension; Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adults patients with chronic respiratory diseases: - 200 adult patients with chronic respiratory diseases will be studied longitudinally and transversely (follow-up: 6 months) in 12 centres.
  1. Sample 1 (n=110 patients) with COPD
  2. Sample 2 (n=30 patients) with Diffuse interstitial lung diseases
  3. Sample 3 (n=30 patients) with Pulmonary Arterial Hypertension primary or secondary (post embolic .....).
  4. Sample 4 (n=30 patients) Adult with Cystic fibrosis
  Interventions: Other: Cross sectional psychometric evaluation of a self-administered dyspnea questionnaire.

INTERVENTIONS:
Other: Cross sectional psychometric evaluation of a self-administered dyspnea questionnaire. — Evaluation will be performed on a group of 200 patients deriving from 4 samples.
  * From these 200 patients, a sub-sample will be evaluated at 7 days (DYSLIM questionnaire only) for reproducibility (n = 50 patients: 10 patients with diffuse interstitial lung disease, 10 patients with cystic fibrosis, 10 patients with arterial pulmonary hypertension, 20 patients with COPD).
  * From these 200 patients, a sub-sample (COPD, n = 60) will be recruited among patients undergoing pulmonary rehabilitation at the beginning of the 6 months separating follow up visit and the initial assessment.
  Other Names: Self-administered dyspnea questionnaire

SUMMARY:
The purpose of this study is the psychometric validation of a self-administered dyspnea questionnaire, usable in clinical practice in order to assess dyspnea and its impact on patients with chronic respiratory diseases.

DETAILED DESCRIPTION:
Dyspnea is a cardinal Respiratory symptom.

According to the ATS dyspnea is the term used to characterize a subjective experience of breathing discomfort, covering qualitatively distinct sensations of varying intensity.

The subjective nature of dyspnea and the high complexity of its determinants explain the often moderate correlations obtained with physiological data. Dyspnea must therefore be measured specifically.

The aim of this study is the cross-sectional and longitudinal psychometric validation of a self-administered dyspnea questionnaire (assessing the impact of dyspnea on activities restriction), usable in clinical practice in order to assess dyspnea and its alterations in adult patients with chronic respiratory diseases.

(COPD, diffuse interstitial lung diseases, Pulmonary arterial hypertension, Cystic fibrosis)

Like any psychometric instrument, an efficient evaluation of dyspnea scale should ideally satisfy all the following required features: evaluative, discriminant, good reproducibility, and high sensitivity to change.

The desired features apart from content validity are reproducibility and especially a high sensitivity to change, particularly following pulmonary rehabilitation.

Thus, this questionnaire should precisely enable to assess the benefit of rehabilitation and it's sustainment in maintenance phase.

ELIGIBILITY:
Inclusion Criteria:

* 1) Sample1: COPD GOLD / ATS > 2 without major co-morbidity

  * Sample 1A: n = 50: group of patients with no change in usual care and no acute event (evaluation of reproducibility)
  * Sample1B: n = 60: patients assessed before and after a qualifying period of pulmonary rehabilitation
* 2) Sample 2 (n = 30): diffuse interstitial lung diseases Criteria: Pulmonary Fibrosis: Idiopathic or nonspecific interstitial lung diseases (NILD) according to international criteria (ATS), sarcoidosis with parenchymal lesions (old classification stage II and III), and exceptionally alveolar proteinosis.
* 3) Sample 3 (n = 30) primary or secondary arterial pulmonary hypertension (post embolic .....).
* 4) Sample4 (n = 30): Adult with Cystic fibrosis.
* 5) patient with stable Status (no exacerbation for at least one month)

Exclusion Criteria:

* 1) Patient under 18 years
* 2) Inability to fill in questionnaires
* 3) Other respiratory disease
* 4) left symptomatic heart failure
* 5) Obesity with a BMI> 35 kg/m2
* 6) Inability to perform PFT (Pulmonary Function Testing)
* 7) Pregnant or breastfeeding woman
* 8) Patient unable to consent
* 9) Lack of social insurance coverage
* 10) Patient in exclusion period because of another protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study Population are adults patients with chronic respiratory diseases (Sample1: COPD; Sample 2: Diffuse interstitial lung diseases; Sample 3: Pulmonary Arterial Hypertension primary or secondary (post embolic .....); Sample 4: Adult with Cystic fibrosis)
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2010-03-16 (Actual); Primary Completion 2014-03-27 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
Psychometric validity of the questionnaire | Until end of treatment (making a total of 6 months)
  Cross-sectional and longitudinal psychometric validation of a self-administered dyspnea questionnaire

SECONDARY OUTCOMES:
Analysis of responses distribution | Until end of treatment (making a total of 6 months)
  Cross-sectional and longitudinal data to assess the psychometric validity of a self-administered dyspnea questionnaire
Structural analysis (in principal components) | Until end of treatment (making a total of 6 months)
  Cross-sectional and longitudinal data to assess the psychometric validity of a self-administered dyspnea questionnaire
External and convergent validity | Until end of treatment (making a total of 6 months)
  Cross-sectional and longitudinal data to assess the psychometric validity of a self-administered dyspnea questionnaire
Internal coherence | Until end of treatment (making a total of 6 months)
  Cross-sectional and longitudinal data to assess the psychometric validity of a self-administered dyspnea questionnaire
Reproducibility | Until end of treatment (making a total of 6 months)
  Cross-sectional and longitudinal data to assess the psychometric validity of a self-administered dyspnea questionnaire
Reproducibility | 7 days
  for a sub sample of 50 patients, Cross-sectional and longitudinal data to assess the psychometric validity of a self-administered dyspnea questionnaire
Discriminating properties | Until end of treatment (making a total of 6 months)
  Cross-sectional and longitudinal data to assess the psychometric validity of a self-administered dyspnea questionnaire
Derivation of a scoring algorithm | Until end of treatment (making a total of 6 months)
  Cross-sectional and longitudinal data to assess the psychometric validity of a self-administered dyspnea questionnaire
Sensitivity to change | Until end of treatment (making a total of 6 months)
  Sensitivity to change will be analyzed in relation to:
  The TDI score, at the Likert scale on changes in dyspnea The scores of quality of life with their respective significant thresholds A the overall medical evaluation A changing EFR parameters with their respective significant thresholds (FEV, DLCO, walk test .....).
  All this are the transversal data necessaries to assess the validation of a psychometric self-administered dyspnea questionnaire.
Minimal difference clinically relevant | Until end of treatment (making a total of 6 months)
  Cross-sectional data necessary to assess the psychometric validity of a self-administered dyspnea questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Perez, MD, Study Chair — CHRU de Lille / Hôpital Calmette - France; Nicolas ROCHE, MD, PhD, Principal Investigator — APHP- Hopital Cochin
Locations (1):
- Service de Pneumologie AP-HP, Hôpitaux Universitaires Paris Centre, Paris, France